CLINICAL TRIAL: NCT03628742
Title: The Use Of Specially Designed Probe Versus Cone- Beam Computerized Tomography In The Measurement Of Gingival Thickness: Diagnostic Accuracy Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Deyaa Darwish, pricipale investigator, Cairo University
Other Study IDs: cairo univesity
Record Dates: First submitted 2018-06-21; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Gingival Thickness; Gingival Biotype; Periodontal Probe
Keywords: periodontal probe; gingival thickness; gingival biotype

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Accurate measurement of gingival thickness is crucial for decision making in the field of Periodontology and implant dentistry. Currently implemented techniques for the detection of gingival biotype are of limited reliability. They possess different drawbacks leading to the necessity for the development of a new method to overcome disadvantages of the available techniques.

the rational of this study is to determine the accuracy of a specially designed probe in comparison to cone- beam computerized tomography which is accurate enough as found by Fu et al 2010.

DETAILED DESCRIPTION:
The success of the esthetic outcome for the anterior teeth restorations and periodontal surgeries depends on several factors such as the gingival biotype, teeth alignment and architecture of the gingiva.

The first who introduced the term biotype are Seibert and Lindhe 1989, they categorized the gingiva to ''thick-flat'' and ''thin-scalloped'' biotypes . Thick biotype is associated with broad tissue and flat gingiva which is also supported by thick bony plate. Thin biotype is associated with thin band of keratinized tissue and scalloped gingiva which is supported by thin bony plate.

A gingival thickness of more or equal to 2 mm is defined as thick biotype and a gingival thickness of less than 1.5 mm as thin biotype. Different gingival biotypes response in different ways to inflammation, restorative and periodontal surgery .

The gingival thickness may predict the outcome of periodontal and restorative treatments. For implant surgery, implant in thin biotype will lead to future peri-implant mucosal recession . The gingival thickness affects the treatment outcome possibly because of the difference in the amount of blood supply of the underlying bone and susceptibility to resorption .

Multiple techniques were proposed to measure the tissue thickness , such as direct measurement ultrasonic devices probe transparency method and cone-beam computed tomography scan

In the direct method, the tissue thickness is measured using a periodontal probe. This method has limitations, such as the angulation of the probe during probing and distortion of tissue during probing

Transgingival method is a simple method to discriminate thin gingival based on the transparency of the periodontal probe through the gingival margin This method was found to be highly reproducible with 85% intra examiner repeatability in a clinical trial of 100 periodontally healthy area . However, this method immeasurable and when presence of pigmented gingiva sometimes hampers the correct identification of gingival biotype .

Another method that was introduced as one of the gingival biotype diagnostic methods is Cone-beam computerized tomography (CBCT), which is widely used to analyze the maxillofacial region . The first who presented commercial CBCT system was Mozzo et al., 1998 . The CBCT offers high-quality diagnostic method and it has become essential in dental practice.

Lascala et al., 2004 have shown the reliability and accuracy when measuring anatomical structures from CBCT images and compared them with measurements of real distances of dry skulls . It was previously reported that CBCT is not indicated for evaluating soft tissue appearance and thickness, and it was considered as a tool for exclusively evaluating hard tissues of the maxillofacial complex . However, recently it has been reported that CBCT can be applied for visualizing and measuring soft tissues of the dento-gingival unit ). Fu et al., 2010 also stated that CBCT provides accurate measurements of both bone and labial soft tissue thickness when compared to caliper method .

A new simple probe is specially designed in an attempt to overcome the angulation problem of the direct method, the complexity and high cost of CBCT and the limitation of the transgingival method.

Aim of Study:

The aim of the study is the evaluation of the use of specially designed probe versus cone- beam computerized tomography in measurement of gingival thickness.

ELIGIBILITY:
Inclusion criteria :

1. In periodontally healthy individuals.
2. Patients with condition indicated for CBCT in upper anterior region
3. Patient age 18-50 years.
4. Intact maxillary central incisors.

Exclusion criteria:

1. Pathological lesion in examined site.
2. Any tooth Malalignment in the examined site.
3. Patients using drugs which may induce gingival enlargement.
4. Pregnant females.
5. Any tooth with any metal restoration in the examined site.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patient will be selected from the Out Patient Clinic from Oral Medicine and Periodontology Department, Faculty of Dentistry Cairo University.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-08-20 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Special Designed Probe | finish the trial in 1 years from the clinical trial registration ( May 2019)
  Assessment of the diagnostic accuracy of Specially designed probe in measuring the gingival thickness in millimeter unit